CLINICAL TRIAL: NCT01069315
Title: Fluid Lavage of Open Wounds (FLOW): A Multi-Center, Blinded, Factorial Pilot Trial Comparing Alternative Irrigating Solutions and Pressures in Patients With Open Fractures
Brief Title: Fluid Lavage of Open Wounds (FLOW): Pilot Trial
Acronym: FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 05-299
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Infection; Wound Healing Problem; Nonunion
Keywords: open wound; solution; pressure; randomized
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal saline and High pressure (Experimental): Irrigation with normal saline delivered at high pressure
  Interventions: Procedure: Type of fluid lavage solution; Procedure: Type of fluid lavage pressure
- Soap solution and High pressure (Experimental): Irrigation with soap solution delivered at high pressure
  Interventions: Procedure: Type of fluid lavage solution; Procedure: Type of fluid lavage pressure
- Normal saline and Low pressure (Experimental): Irrigation with saline solution delivered at low pressure
  Interventions: Procedure: Type of fluid lavage solution; Procedure: Type of fluid lavage pressure
- Soap solution and Low pressure (Experimental): Irrigation with soap solution delivered at low pressure
  Interventions: Procedure: Type of fluid lavage solution; Procedure: Type of fluid lavage pressure

INTERVENTIONS:
Procedure: Type of fluid lavage solution — Comparison of castile soap solution vs. normal saline solution.
Procedure: Type of fluid lavage pressure — Comparison of low pressure vs. high pressure.

SUMMARY:
The purpose of this trial is to investigate whether irrigation solution (soap vs. saline solution), or irrigation pressure (high vs. low) will decrease the rate of infection among patients with open fracture wounds.

DETAILED DESCRIPTION:
Open fractures are an important source of morbidity and are associated with delayed union, nonunion, and infection. Preventing infection through meticulous irrigation and debridement is an important goal in management, and different lavage fluids and irrigation techniques (e.g. high or low pressure lavage) have been described for this purpose. There are, however, a limited number of randomized trials comparing irrigating solutions or irrigating technique. We compared the use of castile soap versus normal saline, as well as high versus low pressure pulsatile lavage on the rates of reoperations and complications in patients with open fracture wounds.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature
* sustained an open fracture of the appendicular skeleton (type I to IIIb).

Exclusion Criteria:

* vascular deficit
* [any] allergy to detergents or castile soap
* previous wound infection or osteomyelitis
* previous fracture with retained hardware in the injured extremity
* operative management more than 24 hours after injury
* use of immunosuppressive medication within six months
* immunological deficiency or disease conditions
* fractures of the hands (distal to the carpus) or toes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, FRCSC, Study Chair — McMaster University; Mohit Bhandari, MD, FRCSC, Principal Investigator — McMaster University; Gordon Guyatt, MD, FRCSC, Principal Investigator — McMaster University; Kyle J Jeray, MD, FRCSC, Principal Investigator — McMaster University
Locations (9):
- United States (3):
  - University of Missouri Health Care, Columbia, Missouri
  - Greenville Hospital System, Greenville, South Carolina
  - East Texas Medical Centre, Tyler, Texas
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Sancheti Institute for Orthopaedics & Rehabilitation, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dormans JP, Fisher RC, Pill SG. Orthopaedics in the developing world: present and future concerns. J Am Acad Orthop Surg. 2001 Sep-Oct;9(5):289-96. doi: 10.5435/00124635-200109000-00002. PMID 11575908
- [Background] Charles Court-Brown, Margaret McQueen, Paul Tornetta III. Trauma. 1st ed. Philadelphia: Lippincott Williams and Wilkins, 2006.
- [Background] Anglen JO. Wound irrigation in musculoskeletal injury. J Am Acad Orthop Surg. 2001 Jul-Aug;9(4):219-26. doi: 10.5435/00124635-200107000-00001. PMID 11476531
- [Background] Khatod M, Botte MJ, Hoyt DB, Meyer RS, Smith JM, Akeson WH. Outcomes in open tibia fractures: relationship between delay in treatment and infection. J Trauma. 2003 Nov;55(5):949-54. doi: 10.1097/01.TA.0000092685.80435.63. PMID 14608171
- [Background] Bhandari M, Guyatt GH, Swiontkowski MF, Schemitsch EH. Treatment of open fractures of the shaft of the tibia. J Bone Joint Surg Br. 2001 Jan;83(1):62-8. doi: 10.1302/0301-620x.83b1.10986. PMID 11245540
- [Background] Bhandari M, Tornetta P 3rd, Sprague S, Najibi S, Petrisor B, Griffith L, Guyatt GH. Predictors of reoperation following operative management of fractures of the tibial shaft. J Orthop Trauma. 2003 May;17(5):353-61. doi: 10.1097/00005131-200305000-00006. PMID 12759640
- [Background] Spencer J, Smith A, Woods D. The effect of time delay on infection in open long-bone fractures: a 5-year prospective audit from a district general hospital. Ann R Coll Surg Engl. 2004 Mar;86(2):108-12. doi: 10.1308/003588404322827491. PMID 15005929
- [Background] Anglen JO. Comparison of soap and antibiotic solutions for irrigation of lower-limb open fracture wounds. A prospective, randomized study. J Bone Joint Surg Am. 2005 Jul;87(7):1415-22. doi: 10.2106/JBJS.D.02615. PMID 15995106
- [Background] Burd T, Christensen GD, Anglen JO, Gainor BJ, Conroy BP, Simpson WA. Sequential irrigation with common detergents: a promising new method for decontaminating orthopedic wounds. Am J Orthop (Belle Mead NJ). 1999 Mar;28(3):156-60. PMID 10195838
- [Background] Petrisor B, Jeray K, Schemitsch E, Hanson B, Sprague S, Sanders D, Bhandari M; FLOW Investigators. Fluid lavage in patients with open fracture wounds (FLOW): an international survey of 984 surgeons. BMC Musculoskelet Disord. 2008 Jan 23;9:7. doi: 10.1186/1471-2474-9-7. PMID 18215287
- [Background] Anglen J, Apostoles PS, Christensen G, Gainor B, Lane J. Removal of surface bacteria by irrigation. J Orthop Res. 1996 Mar;14(2):251-4. doi: 10.1002/jor.1100140213. PMID 8648503
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Brooks R, Rabin RE, de Charro F. The measurement and valuation of health status using EQ-5D: a European perspective. Kluwer Academic Publishers, 2003.
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Background] Owens BD, White DW, Wenke JC. Comparison of irrigation solutions and devices in a contaminated musculoskeletal wound survival model. J Bone Joint Surg Am. 2009 Jan;91(1):92-8. doi: 10.2106/JBJS.G.01566. PMID 19122083
- [Background] Bhandari M, Adili A, Schemitsch EH. The efficacy of low-pressure lavage with different irrigating solutions to remove adherent bacteria from bone. J Bone Joint Surg Am. 2001 Mar;83(3):412-9. doi: 10.2106/00004623-200103000-00014. PMID 11263646
- [Background] Anglen JO, Gainor BJ, Simpson WA, Christensen G. The use of detergent irrigation for musculoskeletal wounds. Int Orthop. 2003;27(1):40-6. doi: 10.1007/s00264-002-0398-5. Epub 2002 Nov 9. PMID 12582808
- [Background] Anglen JO, Apostoles S, Christensen G, Gainor B. The efficacy of various irrigation solutions in removing slime-producing Staphylococcus. J Orthop Trauma. 1994 Oct;8(5):390-6. doi: 10.1097/00005131-199410000-00004. PMID 7996321
- [Background] Malten KE, den Arend JA. Irritant contact dermatitis. Traumiterative and cumulative impairment by cosmetics, climate, and other daily loads. Derm Beruf Umwelt. 1985;33(4):125-32. PMID 4042875
- [Background] Strube DD, Nicoll G. The irritancy of soaps and syndets. Cutis. 1987 Jun;39(6):544-5. PMID 3608584
- [Background] Simion FA, Rhein LD, Morrison BM Jr, Scala DD, Salko DM, Kligman AM, Grove GL. Self-perceived sensory responses to soap and synthetic detergent bars correlate with clinical signs of irritation. J Am Acad Dermatol. 1995 Feb;32(2 Pt 1):205-11. doi: 10.1016/0190-9622(95)90127-2. PMID 7829704
- [Background] Bhandari M, Adili A, Lachowski RJ. High pressure pulsatile lavage of contaminated human tibiae: an in vitro study. J Orthop Trauma. 1998 Sep-Oct;12(7):479-84. doi: 10.1097/00005131-199809000-00009. PMID 9781772
- [Background] Bhandari M, Schemitsch EH, Adili A, Lachowski RJ, Shaughnessy SG. High and low pressure pulsatile lavage of contaminated tibial fractures: an in vitro study of bacterial adherence and bone damage. J Orthop Trauma. 1999 Nov;13(8):526-33. doi: 10.1097/00005131-199911000-00002. PMID 10714777
- [Background] Dirschl DR, Duff GP, Dahners LE, Edin M, Rahn BA, Miclau T. High pressure pulsatile lavage irrigation of intraarticular fractures: effects on fracture healing. J Orthop Trauma. 1998 Sep-Oct;12(7):460-3. doi: 10.1097/00005131-199809000-00005. PMID 9781768
- [Background] Bhandari M, Schemitsch EH. High-pressure irrigation increases adipocyte-like cells at the expense of osteoblasts in vitro. J Bone Joint Surg Br. 2002 Sep;84(7):1054-61. doi: 10.1302/0301-620x.84b7.12532. PMID 12358372
- [Background] Adili A, Bhandari M, Schemitsch EH. The biomechanical effect of high-pressure irrigation on diaphyseal fracture healing in vivo. J Orthop Trauma. 2002 Jul;16(6):413-7. doi: 10.1097/00005131-200207000-00008. PMID 12142830
- [Derived] Sprague S, Tornetta P 3rd, Slobogean GP, O'Hara NN, McKay P, Petrisor B, Jeray KJ, Schemitsch EH, Sanders D, Bhandari M; FLOW Investigators. Are large clinical trials in orthopaedic trauma justified? BMC Musculoskelet Disord. 2018 Apr 20;19(1):124. doi: 10.1186/s12891-018-2029-3. PMID 29678204
- [Derived] FLOW Investigators; Petrisor B, Sun X, Bhandari M, Guyatt G, Jeray KJ, Sprague S, Tanner S, Schemitsch E, Sancheti P, Anglen J, Tornetta P, Bosse M, Liew S, Walter S. Fluid lavage of open wounds (FLOW): a multicenter, blinded, factorial pilot trial comparing alternative irrigating solutions and pressures in patients with open fractures. J Trauma. 2011 Sep;71(3):596-606. doi: 10.1097/TA.0b013e3181f6f2e8. PMID 21378581

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline and High Pressure | Soap Solution and High Pressure | Normal Saline and Low Pressure | Soap Solution and Low Pressure
Started | 27 | 30 | 28 | 26
Completed | 23 | 24 | 23 | 19
Not Completed | 4 | 6 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline and High Pressure | Soap Solution and High Pressure | Normal Saline and Low Pressure | Soap Solution and Low Pressure | Total
Number analyzed (Participants) | 27 | 30 | 28 | 26 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.2) | 39.7 (17.5) | 40.8 (17.8) | 45.3 (18.2) | 42.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9 | 11 | 29
  Male | 25 | 23 | 19 | 15 | 82

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Re-operations (All Subsequent Operative Procedures to Treat an Infection, a Wound Healing Problem, or a Nonunion).
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Soap, Low Pressure | Soap, High Pressure | Saline, Low Pressure | Saline, High Pressure
Number analyzed (Participants) | 26 | 30 | 28 | 27
Participants | 7 | 6 | 3 | 10

2. Secondary Outcome: The Number of Participants With All Operative and Non-operatively Managed Infections, Wound Healing Problems, and Nonunions.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Soap, Low Pressure | Soap, High Pressure | Saline, Low Pressure | Saline, High Pressure
Number analyzed (Participants) | 26 | 30 | 28 | 27
Participants
  Infections treated operatively or nonoperatively | 5 | 8 | 0 | 4
  Nonunion treated operatively or nonoperatively | 2 | 4 | 5 | 8
  Wound healing problem treated operatively or nonop | 5 | 5 | 1 | 9
  No infection, nonunion, or wound healing problems | 14 | 13 | 22 | 6

3. Secondary Outcome: Mean Difference in Health-related Quality of Life and Physical Function From Baseline (Pre-injury) to 12 Months Measured by the SF-12 Questionnaire (Solution).
Description: Solution and pressure were analyzed separately for this outcome. The SF-12 summary scores (PCS-12 and MCS-12) ranges from 0 to 100. Higher scores indicate that a person has better health status, while lower scores indicate poorer health status. Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months per arm.
Time Frame: 1 year
Population: Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months per arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Soap | Saline
Number analyzed (Participants) | 37 | 38
units on a scale
  Mental component summary (MCS) | -1.16 (1.50) | -4.79 (2.30)
  Physical component summary (PCS) | -11.60 (1.32) | -12.49 (1.84)

4. Secondary Outcome: Mean Difference in Health-related Quality of Life and Physical Function From Baseline (Pre-injury) to 12 Months Measured by the EQ-5D Questionnaire (Solution).
Description: Solution and pressure were analyzed separately for this outcome. The EQ-5D summary score ranges from 0 to 1. Higher scores indicate that a person has a better health-related quality of life, while lower scores indicate worse health-related quality of life. Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months per arm.
Time Frame: one year
Population: Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months per arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Soap | Saline
Number analyzed (Participants) | 36 | 39
units on a scale | -0.14 (0.33) | -0.19 (0.33)

5. Secondary Outcome: Mean Difference in Health-related Quality of Life and Physical Function From Baseline (Pre-injury) to 12 Months Measured by the SF-12 Questionnaire (Pressure)
Description: as for outcome 3
Time Frame: one year
Population: Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months per arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 38 | 37
units on a scale
  Mental component summary (MCS) | -12.16 (1.84) | -11.94 (1.95)
  Physical component summary (PCS) | -4.59 (1.97) | -1.37 (2.28)

6. Secondary Outcome: Mean Difference in Health-related Quality of Life and Physical Function From Baseline (Pre-injury) to 12 Months Measured by the EQ-5D Questionnaire (Pressure)
Description: Solution and pressure were analyzed separately for this outcome. The EQ-5D summary score ranges from 0 to 1. Higher scores indicate that a person has a better health-related quality of life, while lower scores indicate worse health-related quality of life. Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months.
Time Frame: one year
Population: Please note that the values reported are mean differences in scores from baseline (pre-injury) to 12 months per arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Pressure | Low Pressure
Number analyzed (Participants) | 40 | 35
units on a scale | -0.18 (0.033) | -0.15 (0.033)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Events were monitored/ assessed in such a manner that the specific Adverse Event Terms cannot be separated
Arm/Group | Soap, Low Pressure | Soap, High Pressure | Saline, Low Pressure | Saline, High Pressure
Serious Adverse Events (participants affected / at risk) | 13/27 | 14/30 | 9/26 | 11/27
Other Adverse Events (participants affected / at risk) | 4/27 | 8/30 | 0/26 | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soap, Low Pressure (N=27) | Soap, High Pressure (N=30) | Saline, Low Pressure (N=26) | Saline, High Pressure (N=27)
All SAEs (Surgical and medical procedures) | 13 (25) | 14 (26) | 9 (15) | 11 (31)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soap, Low Pressure (N=27) | Soap, High Pressure (N=30) | Saline, Low Pressure (N=26) | Saline, High Pressure (N=27)
All other AEs (Surgical and medical procedures) | 4 (4) | 8 (12) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No